CLINICAL TRIAL: NCT03699371
Title: Influence of Early vs Late Supplemental ParenteraL Nutrition on Long-term Quality of Life in ICU Patients After Gastrointestinal Oncological Surgery. A Prospective, Randomised, Multi-centre Assessor-blinded Study. hELPLiNe Trial
Brief Title: Influence of Early vs Late SPN on Long-term Quality of Life in ICU Patients After Gastrointestinal Oncological Surgery
Acronym: hELPLiNe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Lublin (Other)
Collaborators: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Paweł Piwowarczyk, Principal Investigator, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KE-0254/152/2018
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Nutrition Aspect of Cancer
Keywords: early parenteral nutrition; supplemental nutrition; quality of life; oncological surgery; critical care
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Intervention Model Description: prospective, randomised, multi-centre assessor-blinded study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Supplemental Parenteral Nutrition (Experimental): Intervention group: would receive EN reaching up to 20 % of daily nutritional requirements and early (on first day of stay in ICU) provision (of up to 80%) of protein (2 g/kg/ day or in case of continuous renal replacement therapy (CRRT) 2,5 g/kg/ day) and caloric (15-20 kcal/kg/day) needs in SPN that would be continued until 7th day of stay in ICU for the purpose of the study.
  Interventions: Procedure: Early Supplemental Parenteral Nutrition
- Late Supplemental Parenteral Nutrition (No Intervention): Control group: would receive EN reaching up to 20 % of daily nutritional requirements and late (of up to 80%) of protein (2 g/kg/ day or in case of CRRT 2,5 g/kg/ day) and caloric (15-20 kcal/kg/day ) in SPN on 7th day of stay in ICU if it is not already met via enteral route.

INTERVENTIONS:
Procedure: Early Supplemental Parenteral Nutrition — Intervention group: would receive EN reaching up to 20 % of daily nutritional requirements and early (on first day of stay in ICU) provision (of up to 80%) of protein (2 g/kg/ day or in case of CRRT 2,5 g/kg/ day) and caloric (15-20 kcal/kg/day) needs in SPN that would be continued until 7th day of stay in ICU. Central venous catheter placement would not be assessed as a part of intervention due to the fact that it is a part of routine medical activities performed during admission to ICU.
  Arms: Early Supplemental Parenteral Nutrition

SUMMARY:
BACKGROUND: Nutrition plays a significant role in ICU treatment, and may influence mortality and length of stay in ICU. Enteral route (EN) is preferential to parenteral route (PN) in provision of daily nutritional requirements. When enteral route is insufficient, supplemental parenteral nutrition (SPN) is recommended. Optimal timing of SPN in acute phase of illness remains elusive. ICU patients suffer significant lean body mass loss, in majority, in the first 7-10 days of stay. Optimal provision of protein may prevent muscle wasting. Lean body mass is essential for optimal physical functioning after treatment. Although ICU mortality has been reduced lately, the number of patients going to rehabilitation after ICU stay has tripled. Patients after oncological surgery of the gastrointestinal tract may be threatened with impairment of physical functioning after ICU treatment.

AIM: To compare the influence of early and late supplemental parenteral nutrition on long-term physical functioning in ICU patients after oncological surgery of the gastrointestinal tract.

STUDY DESIGN: Prospective, randomised, multi-centre assessor-blinded study. METHODS & ANALYSIS: Patients will be randomised into intervention group that would receive SPN on first day, and would be continued until 7th day of stay in ICU. Control group would receive SPN on 7th day of stay in ICU, when it is not then already met via enteral route. Physical Component of SF-36 Scale at 6 month after ICU admission will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. ICU patients in the acute phase of critical illness after gastrointestinal oncological surgery.
2. Admitted to the ICU during the previous 24 hours with a minimum expected ICU stay of ≥5 days
3. Central venous access available for continuous infusion of the study drugs
4. Sequential Organ Failure Assessment (SOFA) score ≥2
5. Written informed consent from the patient or the patient's legal representative

Exclusion Criteria:

Contraindication against SPN or inability to receive SPN via central venous access

1. Received PN within 7 days before randomisation
2. Expected to receive ≥20% of energy via supplemental enteral nutrition (EN) and/or non-nutritional sources (e.g. glucose solution for drug dilution or lipids from propofol) during the first 3 nutritional treatment days
3. Inability to initiate EN prior to randomization
4. Body mass index (BMI) <17 kg/m2 or >35 kg/m2
5. Any severe, persistent blood coagulation disorder with uncontrolled bleeding
6. Any congenital errors of amino acid metabolism
7. Known hypersensitivity to fish, egg, soybean proteins, peanut proteins, or to any of the active substances or excipients contained in SPN.
8. Known hypersensitivity to milk protein or to any other substance contained in SPN
9. Acute liver failure with encephalopathy, including intoxication (e.g. paracetamol, death cap, golden chain) and/or liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma glutamyl transferase [GGT]) or bilirubin exceeding 10 x ULN
10. Hemophagocytic syndrome
11. Known history of human immunodeficiency virus (HIV), hepatitis B and/or C
12. Pregnancy or lactation
13. Patient unlikely to survive to 6 months due to underlying illness
14. Receiving end-of-life-care

    Laboratory Exclusions:
15. Hypertriglyceridemia characterised by serum triglyceride levels >4 mmol/L [>350 mg/dL])
16. Treatment-refractory, clinically significant major abnormality in the serum concentration of any electrolyte (sodium, potassium, magnesium, total calcium, chloride, inorganic phosphate)

    Concomitant Therapy Exclusions:
17. Chronic maintenance therapy with systemic glucocorticoid steroids (Hydrocortisone >0.3 mg/kg/d)
18. Concomitant administration of chemotherapy
19. Administration of growth hormone and teduglutide within the previous 4 weeks

    Other Exclusions:
20. Chronic liver failure ( Child -Pugh scale B or C) e.g. secondary to drug or alcohol abuse
21. Participation in another interventional clinical trial within the previous 4 weeks
22. Previous inclusion in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Long-term quality of life at 3 months | Physical component of 36 -SF questionnaire at 3 months after admission to ICU
  Long-term quality of life measured in physical component of 36 -SF questionnaire
Long-term quality of life at 6 months | Physical component of 36 -SF questionnaire at 6 months after admission to ICU
  Long-term quality of life measured in physical component of 36 -SF questionnaire

SECONDARY OUTCOMES:
Enteral route intolerance | At day 3 since admission to ICU
  Inability to administer up to 60% of protein needs on 3rd day via enteral route
Thickness of diaphragm | 1st, 3rd, 5th day of ICU stay
  Change from baseline in ultrasound measured thickness of diaphragm
Protein delivery | For 7 days since admission to ICU
  Protein delivery defined as daily input of proteins via SPN
Energy Intake | For 7 days since admission to ICU
  Energy delivery defined as daily input of calories via SPN
Insulin dose | For 7 days since admission to ICU
  Insulin dose defined as summary daily input of insulin
Blood glucose profile | For 7 days since admission to ICU
  Blood glucose profile defined as mean daily glucose level
Organic phosphorus level | For 7 days since admission to ICU
  Organic phosphorus level defined as result in blood test performed daily
Sequential Organ Failure Assessment score ( SOFA score) | For 28 days since admission to ICU or till discharge
  We will collect data regarding changes from baseline SOFA score - to determine the extent of a person's organ function failure. SOFA scoring system is useful in predicting the clinical outcomes of critically ill patients. Patient can be scored from 0 to 24. If the patient is scored 0 than the patient is in a good state and predicted mortality is low, while 24 is the worst result with expected very high mortality rate.
Mechanical Ventilation | For 28 days since admission to ICU or till discharge
  Numbers of days of mechanical ventilation
Length of stay in the ICU | For 28 days since admission to ICU or till discharge
  Numbers of days of patient stay in ICU
ICU mortality | For 28 days since admission to ICU or till discharge
Hospital mortality | For 28 days since admission to ICU or till discharge
Length of stay in hospital | For 28 days since admission to ICU or till discharge
  Numbers of days of patient stay in hospital
Health-care associated infection | For 28 days since admission to ICU or till discharge
  New onset of health-care associated infection
Antibiotic-free days | For 28 days since admission to ICU or till discharge
  Number of days patient was not given the antibiotics

OTHER OUTCOMES:
PCS SF-36 change | From enrollment till 6 months assessment
  Change from baseline in PCS SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Piwowarczyk, MD PhD, Principal Investigator — Medical University in Lublin
Locations (2):
- Poland (2):
  - 2nd Department of Anesthesiology and Critical Care, Medical University of Lublin, Lublin, Lublin Voivodeship
  - Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicolo M, Heyland DK, Chittams J, Sammarco T, Compher C. Clinical Outcomes Related to Protein Delivery in a Critically Ill Population: A Multicenter, Multinational Observation Study. JPEN J Parenter Enteral Nutr. 2016 Jan;40(1):45-51. doi: 10.1177/0148607115583675. Epub 2015 Apr 21. PMID 25900319
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Sundstrom Rehal M, Liebau F, Tjader I, Norberg A, Rooyackers O, Wernerman J. A supplemental intravenous amino acid infusion sustains a positive protein balance for 24 hours in critically ill patients. Crit Care. 2017 Dec 6;21(1):298. doi: 10.1186/s13054-017-1892-x. PMID 29212550
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] Allingstrup MJ, Kondrup J, Wiis J, Claudius C, Pedersen UG, Hein-Rasmussen R, Bjerregaard MR, Steensen M, Jensen TH, Lange T, Madsen MB, Moller MH, Perner A. Early goal-directed nutrition versus standard of care in adult intensive care patients: the single-centre, randomised, outcome assessor-blinded EAT-ICU trial. Intensive Care Med. 2017 Nov;43(11):1637-1647. doi: 10.1007/s00134-017-4880-3. Epub 2017 Sep 22. PMID 28936712
- [Background] Reignier J, Boisrame-Helms J, Brisard L, Lascarrou JB, Ait Hssain A, Anguel N, Argaud L, Asehnoune K, Asfar P, Bellec F, Botoc V, Bretagnol A, Bui HN, Canet E, Da Silva D, Darmon M, Das V, Devaquet J, Djibre M, Ganster F, Garrouste-Orgeas M, Gaudry S, Gontier O, Guerin C, Guidet B, Guitton C, Herbrecht JE, Lacherade JC, Letocart P, Martino F, Maxime V, Mercier E, Mira JP, Nseir S, Piton G, Quenot JP, Richecoeur J, Rigaud JP, Robert R, Rolin N, Schwebel C, Sirodot M, Tinturier F, Thevenin D, Giraudeau B, Le Gouge A; NUTRIREA-2 Trial Investigators; Clinical Research in Intensive Care and Sepsis (CRICS) group. Enteral versus parenteral early nutrition in ventilated adults with shock: a randomised, controlled, multicentre, open-label, parallel-group study (NUTRIREA-2). Lancet. 2018 Jan 13;391(10116):133-143. doi: 10.1016/S0140-6736(17)32146-3. Epub 2017 Nov 8. PMID 29128300
- [Derived] Piwowarczyk P, Kutnik P, Borys M, Rypulak E, Potrec-Studzinska B, Sysiak-Slawecka J, Czarnik T, Czuczwar M. Influence of Early versus Late supplemental ParenteraL Nutrition on long-term quality of life in ICU patients after gastrointestinal oncological surgery (hELPLiNe): study protocol for a randomized controlled trial. Trials. 2019 Dec 27;20(1):777. doi: 10.1186/s13063-019-3796-3. PMID 31881984